CLINICAL TRIAL: NCT04254237
Title: Trocar Site Hernia After Laparoscopic Cholecystectomy: Randomized Clinical Trial Comparing Supra Versus Infraumbilical Incision for Umbilical Trocar Entry
Brief Title: Trocar Site Hernia After Laparoscopic Cholecystectomy, Supra Versus Infraumbilical Incision for Umbilical Trocar Entry
Acronym: HOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Hospitalario La Mancha Centro (Other)
Responsible Party: Principal Investigator, Antonio Morandeira Rivas, MD PhD, General Surgeon and Residency program director, Complejo Hospitalario La Mancha Centro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 99-B
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Incisional Hernia; Cholecystectomy, Laparoscopic
Keywords: Trocar site hernia; Laparoscopy; Laparoscopic cholecystectomy; Minimally invasive surgery
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Infraumbilical Hasson trocar incision.
  Interventions: Procedure: Infraumbilical Hasson trocar incision
- Control group (Sham Comparator): Supraumbilical Hasson trocar incision.
  Interventions: Procedure: Supraumbilical Hasson trocar incision

INTERVENTIONS:
Procedure: Infraumbilical Hasson trocar incision — Infraumbilical Hasson trocar incision
  Arms: Intervention group
Procedure: Supraumbilical Hasson trocar incision — Supraumbilical Hasson trocar incision
  Arms: Control group

SUMMARY:
Trocar site hernia is a specific complication of laparoscopic surgery. The increasingly frequent use of the laparoscopic approach has resulted in an increase in the number of hernias, mainly at the umbilical area. The appearance of a trocar site hernia can cause complications in the short and long term to the patient who may end up needing a reoperation.

In this study we want to compare the supraumbilical versus the infraumbilical location of the laparoscopy entry trocar, in terms of incisional hernia incidence.

DETAILED DESCRIPTION:
Trocar site hernias have been considered as an underestimated problem by some surgeons. It's incidence varies in the literature between studies, which may be related to an insufficient diagnosis due to poor clinical manifestation and / or the lack of long-term follow-up of patients in some studies.

There are many risk factors that have been related to the trocar site hernia development. On one side, the patient clinical factors as the age, presence of obesity, diabetes mellitus or the smoking habits. On the other side, some risk factors related to the surgical technique have been described, as the entry technique, the size and the locations of the trocars, the fascial closure, the duration of the surgery or the infection of the surgical wound.

Regarding the location of the trocars, it seems that the middle line has more risk of incisional hernia than the lateral areas in the abdomen. However, the trocar locations out of the middle line is not always possible, especially in certain surgeries as the laparoscopic cholecystectomy where it can be necessary an expansion of the incision for removing the specimen. In the concrete case of laparoscopic cholecystectomy, the belly is usually the most popular region for placing the first trocar. However, there is not much evidence about the influence of the most popular locations of the umbilical trocar incision (supra or infraumbilical) in the development of incisional hernias.

In the middle line, the infraumbilical region presents a great ability to adapt to pressure changes, as it physiologically occurs during the pregnancy. On the other side, while the primary hernias in the supraumbilical and umbilical region are common, these are not produced in the infraumbilical region. Besides, in anatomical studies of the linea alba, a higher thickness of the fibres in the infraumbilical region has been observed, along with a different spatial arrangement, predominating the transverse fibres in the infraumbilical region and the oblique ones in the supraumbilical region. Therefore, we hypothesize whether the infraumbilical location of the trocar in the midline, theoretically a more protected region, can reduce the incidence of trocar site hernia in our patients.

The aim of this study is to compare the incidence of the Hasson trocar site hernia between the supra and infraumbilical locations a year after surgery, in high risk patients for trocar site hernia subjected to elective laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Ability to understand the trial information.
* Patients with symptomatic gallstones or polyps scheduled for laparoscopic cholecystectomy.
* Elective surgery.
* One year potential follow-up.
* Patients that experience one or more of the following Trocar Site Hernia risk factors:

  * Over 60 years old.
  * Obesity, defined as Body Mass Index (BMI) > 30 Kg/m2.
  * Diabetes mellitus (DM).
  * Bronchopathy: A diagnosed Chronic Obstructive Pulmonary Disease (COPD) or smokers of more than 25 cigarette packages/year.
* Accept to participate in the study and sign the informed consent.

Exclusion Criteria:

* Contraindication to conduct a laparoscopic cholecystectomy.
* Patients with previous open supramesocolic surgery.
* Patients with previous surgery that affects the umbilical region.
* Patients with umbilical hernia or history of umbilical hernia surgical correction.
* A greater than 30 cm xifo-umbilical distance.
* Extreme obesity (Body Mass Index > 50 kg/m2).
* Cancer patients or in immunosuppressive therapy.
* Connective tissue disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Trocar site hernia | One year
  Number of patients presenting a trocar site hernia, at the periumbilical incision, one year after laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
Umbilical wound complications different from Trocar Site Hernia | 24 hours, 7 days, 30 days, 6 months and 1 year.
  Infection, seroma or ecchymosis at the umbilical wound
Non-umbilical wounds complications | 24 hours, 7 days, 30 days, 6 months and 1 year.
  Hernia, infection, seroma, ecchymosis or evisceration at non-umbilical wounds.
Other complications | 24 hours, 7 days, 30 days, 6 months and 1 year.
  Other complications not related to the surgical wound
Surgical time | Day 0
  Measured in minutes from the first incision until the complete closure of the last surgical wound
Conversion | Day 0
  Conversion rate to open surgery (yes/no).
Hospital stay | Day 0
  Measured in hours from the surgery to the patient discharge.
Postoperative pain | 24 hours and 7 days after surgery.
  Measured using the Visual Analogue Scale (VAS), with a punctuation between 0 (no pain) and 10 (the worst conceivable pain).
Perceived Quality of Life | baseline, one month and a year after surgery.
  Measured using the SF-36 questionnaire,
Aesthetic result | Six months and a year of the surgery.
  Measured using the Visual Analogue Scale, with a punctuation between 0 (not at all satisfied) and 10 (maximum satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Morandeira-Rivas, MD PhD, Principal Investigator — La Mancha Centro General Hospital; Carlos Moreno Sanz, MD PhD FACS, Study Chair — La Mancha Centro General Hospital
Locations (3):
- Spain (3):
  - La Mancha Centro General Hospital, Alcázar de San Juan, Ciudad Real
  - Tomelloso General Hospital, Tomelloso, Ciudad Real
  - Valdepeñas General Hospital, Valdepeñas, Ciudad Real